CLINICAL TRIAL: NCT04430920
Title: Blood Pressure Management on Cardiovascular AdveRse Events After Major Abdominal Surgery (BP-CARES): A Randomized Controlled Trial
Brief Title: Blood Pressure Management on Cardiovascular AdveRse Events After Major Abdominal Surgery
Acronym: BP-CARES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Xinqiao Hospital of Chongqing (Other); Henan Provincial People's Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NFEC-2019-261
Record Dates: First submitted 2020-06-11; First posted 2020-06-16 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Cardiovascular Complication
Keywords: Intraoperative blood pressure; Major abdominal surgery; Cardiovascular complication

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive intraoperative blood pressure management (Active Comparator)
  Interventions: Other: Intensive intraoperative blood pressure management
- Conventional intraoperative blood pressure management (Placebo Comparator)
  Interventions: Other: Conventional intraoperative blood pressure management

INTERVENTIONS:
Other: Intensive intraoperative blood pressure management — Targeting intraoperative mean arterial pressure ≥ 80 mmHg.
  Arms: Intensive intraoperative blood pressure management
Other: Conventional intraoperative blood pressure management — Targeting intraoperative mean arterial pressure ≥ 65 mmHg or 60% of the baseline level (use the higher target).
  Arms: Conventional intraoperative blood pressure management

SUMMARY:
This study is a multicenter randomized controlled trial comparing an intensive intraoperative blood pressure management strategy versus conventional practice for preventing cardiovascular events in high-risk patients undergoing major abdominal surgery.

DETAILED DESCRIPTION:
Intraoperative hypotension has been associated with cardiovascular events after non-cardiac surgery. However, whether avoiding intraoperative hypotension can reduce the incidence of postoperative cardiovascular events remains unclear. The objective of this study is to assess the effects of an intensive intraoperative blood pressure management strategy (to maintain intraoperative MAP ≥ 80mmHg) with that of conventional practice (to maintain intraoperative MAP ≥ 65mmHg) on the incidence of cardiovascular events after major abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 45 years;
2. Undergoing major abdominal surgery under general anesthesia (expected surgery time >2h, expected length of postoperative stay >2d);
3. Fulfill ≥1 of the following criteria (a-f): a. history of coronary artery disease; b. history of stroke; c. history of peripheral arterial disease; d. history of congestive heart failure; e. preoperative NT-proBNP >200 pg/mL or BNP >92 mg/L f. preoperative troponin > upper limit of normal; or fulfill ≥2 of the following criteria (g-l); g. history of chronic kidney disease (preoperative sCr >133μmol/L or 1.5 mg/dL); h. diabetes requiring medical treatment; i. smoking in the past >2 years; j.≥ 65 years of age; k. hypertension requiring medical treatment l. history of hypercholesterolemia.

Exclusion Criteria:

1. ASA score ≥5;
2. Severe untreated or uncontrolled hypertension (preoperative SBP>180mmHg and/or DBP>110mmHg);
3. End-stage renal disease requiring renal-replacement therapy;
4. Acute cardiovascular event within 1 month of surgery, including acute heart failure, acute coronary syndrome and stroke;
5. Preoperative sepsis or septic shock;
6. Preoperative requirement of vasopressor infusion;
7. Current participation in another interventional study;
8. Previous participation in this study;
9. Pregnant or breastfeeding women.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2022-09-23 (Actual); Study Completion 2025-04-08 (Actual)

PRIMARY OUTCOMES:
Number of participants with major adverse cardiac events | 30-day after surgery
  A composite of myocardial injury/infarction, new-onset clinically important arrhythmia, heart failure, stroke, cardiac arrest, and all-cause death after surgery

SECONDARY OUTCOMES:
Number of participants with non-cardiovascular complications | 30-day after surgery
  Postoperative acute kidney injury, infection, pulmonary complications, delirium, gastrointestinal complications (GI infarction, bleeding, perforation, obstruction), venous thromboembolism, anastomotic fistula, bleed requiring transfusion
Days alive and at home | 30-day after surgery
Number of participants who died or developed disability | 180-day after surgery
  Disability is assessed based on 12-item WHO Disability Assessment Schedule (WHODAS 2.0)

OTHER OUTCOMES:
For patients receiving radical cancer resection: overall survival | 3-year after surgery
For patients receiving radical cancer resection: disease-free survival | 3-year after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Bingcheng Zhao, MD, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (3):
- China (3):
  - Xinqiao Hospital of Chongqing, Chongqing, Chongqing Municipality
  - Southern Medical University Nanfang Hospital, Guangzhou
  - Henan Provincial People's Hospital, Zhengzhou

IPD SHARING:
Plan to Share IPD: Yes
The deidentified IPD will be shared upon reasonable request after study completion.